CLINICAL TRIAL: NCT05801926
Title: Promoting BEST (BEtter, Faster, Longer, STronger) Walking for People With Parkinson's
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Nancy Mayo (Other)
Collaborators: MedTeq (Industry); Healthy Brains for Healthy Lives (Unknown); Mitacs (Industry); PhysioBiometrics Inc. (Unknown)
Responsible Party: Sponsor-Investigator, Nancy Mayo, James McGill Professor, McGill University
Organization: McGill University (Other)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: A00-B37-22A / eRAP 22-04-037
Record Dates: First submitted 2023-02-04; First posted 2023-04-06 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-03

CONDITIONS: Parkinson Disease
Keywords: gait; walking; wearable; feedback; motivation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Individual, blocked, stepped-wedge
Masking Description: Everyone eventually gets the intervention, it is the order that is randomized. The outcome is gait quality measured directly from the sensor and is not affected by observers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate assignment (Experimental): Within this block, half are assigned to receive the sensor right away.
  Interventions: Device: Heel2Toe[TM] sensor
- Delayed assignment (Active Comparator): Within this block, half are assigned to receive the sensor after a delay of 3 to 4 weeks
  Interventions: Device: Heel2Toe[TM] sensor

INTERVENTIONS:
Device: Heel2Toe[TM] sensor — Heel2Toe is a new generation of wearables that provides real-time auditory feedback when the person takes a good step, one in which the step is initiated with a strong heel strike.

SUMMARY:
This project aims to improve how people with Parkinson's Disease (PD) walk. The global aim is to identify obstacles and solutions for people with PD for adopting technology to track and improve their gait to make them better and safer walkers. To meet this aim members of Parkinson Quebec will be surveyed about their technology readiness, physical, cognitive, and psychological health, and rehabilitation access. The survey should not take more than 20 minutes to complete on the web. Subsequently, a random sample of 100 survey participants will be offered a wearable device, the Heel2ToeTM sensor, designed to improve gait quality. This device emits a beep when a proper step is taken. This external cue reinforces the adoption of an adequate gait. In addition to the device, participants will be offered 5 sessions of telemonitoring to help them use the device optimally. Monitoring of use and outcomes will be over 3 months and the sensor is theirs to keep.

DETAILED DESCRIPTION:
The global aim of this research program is to identify technical, attitudinal, and motivational obstacles and solutions for people with PD for adopting technology to improve gait and to quantify changes in gait biomechanics that will make participants better and safer walkers, ultimately improving physical function, physical activity, motivation, and quality of life.

Specific objective: Among members of the PQ who meet the criteria for technology readiness and have sufficient walking capacity to use the Heel2ToeTM sensor at home, the objectives are to estimate the extent to which they: (1) require support from the technology and rehabilitation team to optimize use; (2) use the sensor; (3) and change gait pattern, walking behaviours, motivation and functional and quality of life indicators over a period of 3 months.

Design: An individualized, blocked, stepped-wedge design will be used, a design favoured for implementation science questions 63,64 and applicable here as the team does not have the resources to implement the technology to all participants all at once. Parkinson Quebec has provided funds to provide sensors for 100 people. Variable size clusters of people will be formed and randomized to receive the Heel2Toe sensor, training, and remote supervised use, at intervals of 3 weeks. The cluster size will be randomly determined ranging from 4 to 10. As everyone selected for the implementation have already filled out the survey, there is a common data set at project entry. This assessment will be repeated prior to being entered into the Heel2Toe phase and then 3 months later.

ELIGIBILITY:
Inclusion Criteria:

Technology readiness will be determined by the following criteria:

* has wifi
* has a smartphone that is recent enough to support the technology or willing to acquire one
* uses apps on the smartphone on most days of the week with or without the aid of another person
* positively endorses the question "Are you interested in learning new things?"58 and "I walk outdoors on most days, weather permitting."

To screen participants for their capacity to use the Heel2Toe sensor, participants meeting the technology readiness criteria will be instructed to send a smartphone video of themselves doing a modified Timed-up-an-Go test65 in which the person, stands up from a chair, walks minimum of 10 meters (original TUG is 3 m.), turns, walks back to the chair, and sits down (long-TUG).

Exclusion Criteria:

* unable to do the long TUG without assistance or need for a walking aid
* unable to recover balance independently from a perturbation during execution of the long TUG
* unable to reinitiate movement without assistance or without losing balance during a freezing event occurring during the long TUG. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-01-31 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Angular velocity of ankle at heel strike averaged over a walk of a least 50 steps | Change from baseline to 3 months, 6 months, 1 year
  degrees per second
Angular velocity of ankle during push-off averaged over a walk of a least 50 steps | Change from baseline to 3 months, 6 months, 1 year
  degrees per second
Angular velocity of ankle during foot swing averaged over a walk of a least 50 steps | Change from baseline to 3 months, 6 months, 1 year
  degrees per second
Co-efficient of variation of angular velocity of ankle during three phases of gait cycle, heel-strike, push-off, swing averaged over a walk of at least 50 steps | Change from baseline to 3 months, 6 months, 1 year
  ratio of standard deviation to mean converted to percent.

SECONDARY OUTCOMES:
Motivation | Change from baseline to 3 months, 6 months, 1 year
  Starkstein Apathy Scale (0-42, higher worse)
Apathy | Change from baseline to 3 months, 6 months, 1 year
  Motivation Inventory (0-68, higher worse)
Walking behaviour | Change from baseline to 3 months, 6 months, 1 year
  Daily step count
Health-related quality of life (HRQL) | Change from baseline to 3 months, 6 months, 1 year
  EQ-5D-5L (0-1; higher is better)
Health-related quality of life (HRQL)better) | Change from baseline to 3 months, 6 months, 1 year
  Preference-based Parkinson Index (0-100; higher is better)
Self-reported Cognitive Ability | Change from baseline to 3 months, 6 months, 1 year
  Communicating Cognitive Concerns (C3Q: 0-36, higher is better)
Cognitive Performance Test | Change from baseline to 3 months, 6 months, 1 year
  Symbol Digit Modality Test (errors in 90 seconds)

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Division of Clinical Epidemiology, Montreal, Quebec
  - Research Institute of the McGill University Health Center, CORE, 5252 de Maisonneuve, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No